A falls prevention programme to improve quality of life, physical function and falls efficacy in older people receiving home help services: Study protocol for a randomised controlled trial

Last updated: 06/23-2017

#### **Authors:**

Maria Bjerk (Corresponding author) Faculty of Health Sciences Oslo and Akershus University College PO Box 4 St. Olavs plass 0130 Oslo, Norway

maria.bjerk@hioa.no +47 67 23 66 83

Therese Brovold
Faculty of Health Sciences
Oslo and Akershus University College
therese.brovold@hioa.no

Dawn A Skelton Institute of Applied Health Research School of Health and Life Sciences, Glasgow Caledonian University, UK dawn.skelton@gcu.ac.uk

Astrid Bergland Faculty of Health Sciences Oslo and Akershus University College astrid.bergland@hioa.no

Published under the terms of the CC BY 4.0 licence: Bjerk M, Brovold T, Skelton DA, Bergland A: **A** falls prevention programme to improve quality of life, physical function and falls efficacy in older people receiving home help services: study protocol for a randomised controlled trial. *BMC Health Services Research* 2017, **17**(1): 559. DOI: 10.1186/s12913-017-2516-5

A falls prevention programme to improve quality of life, physical function and falls efficacy in older people receiving home help services: Study protocol for a randomised controlled trial

### **Abstract**

### **Background:**

Falls and fall-related injuries in older adults are associated with great burdens, both for the individuals, the health care system and the society. Previous research has shown evidence for the efficiency of exercise as falls prevention. An understudied group are older adults receiving home help services, and the effect of a falls prevention programme on health-related quality of life is unclear. The primary aim of this randomised controlled trial is to examine the effect of a falls prevention programme on quality of life, physical function and falls efficacy in older adults receiving home help services. A secondary aim is to explore the mediating factors between falls prevention and health-related quality of life.

#### Methods:

The study is a single-blinded randomised controlled trial. Participants are older adults, aged 67 or older, receiving home help services, who are able to walk with or without walking aids, who have experienced at least one fall during the last twelve months and who have a Mini Mental State Examination of 23 or above. The intervention group receives a programme, based on the Otago Exercise Programme, lasting twelve weeks including home visits and motivational telephone calls. The control group receives usual care. The primary outcome is health-related quality of life (SF-36). Secondary outcomes are leg strength, balance, walking speed, walking habits, activities of daily living, nutritional status and falls efficacy. All measurements are performed at baseline, following intervention at three months and at six months' follow-up. Sample size, based on the primary outcome, is set to 150 participants randomised into the two arms, including an estimated 15-20% drop out. Participants are recruited from six municipalities in Norway.

#### **Discussion:**

This trial will generate new knowledge on the effects of an exercise falls prevention programme among older fallers receiving home help services. This knowledge will be useful for clinicians, for health managers in the primary health care service and for policy makers.

**Trial registration:** ClinicalTrials.gov. NCT02374307. First registration, 16/02/2015.

**Keywords:** Falls prevention, Home help services, Elderly, Quality of life, Older adults, Exercise, Balance, Preventative care

# Background

# Older adults and health-related quality of life

Health-related quality of life (HRQOL) is of great interest, both with respect to individuals themselves as well as a primary concern of public health administrations and professionals. The remarkable increase in life expectancy in the twentieth century implies a need to focus on factors capable of promoting a high level of HRQOL into old age. In fact, older adults seem to prefer a high HRQOL more than longevity, and researchers have concluded that the key challenge is to preserve a high level of HRQOL rather than increase length of life [1, 2]. HRQOL is a subjective, multidimensional concept shaped by, but not entirely dependent upon, the effects of disease and treatment [3]. The WHO Quality of life (QOL) group defines QOL as "individuals' perception of their position in life in the context of the culture and value systems in which they live, and in relation to their goals, expectations, standards and concerns" [4]. Public health policies in many European countries are therefore primarily concerned with keeping older people living independently in the community with a good quality of life [5-7]. The raise in number of older adults implies more people with chronic diseases and a greater challenge for the health care system in finding effective and feasible interventions to reach this goal [5-8].

Aiming to enable older people to live at home as long as possible, the municipalities in Norway are responsible for providing services in the form of home help for older people [9]. Home help includes services that assist instrumental activities of daily living (iADL), such as vacuum cleaning, and personal activities of daily living (pADL), such as getting dressed, safety alarm services to provide assistance if they fall, and social support. The most important predictor of home care use seems to be dependency in IADL and ADL and cognitive impairment [10]. Home help receivers constitute a transitional group between independent community living older people, and people living in residential care facilities/nursing homes [11]. The combination of the increase of older people and the use of the so-called LEON ("lowest most efficient level of care") principle [6], makes this a steadily growing group in society, and can be seen as an especially vulnerable group among the older population. Moreover, as economic resources are scarce, there seems to be more focus on post-acute care instead of health promotion and prevention to maintain older adults at home [12]. To date there is no evidence-based practice standard for falls-prevention in Norwegian home care services.

# Older adults and falls

Falls and fall-related injuries are common in older adults and are associated with substantial economic costs that are borne by individuals, the community, and the medical system as a whole [13, 14]. Up to 40% of all nursing home admissions have been found to relate to falls and instability [15]. Important risk factors for falling in the group of older adults are impaired balance and gait, polypharmacy and a history of falls [16]. Poor nutritional status has also been associated with an increased risk of falling, [17] and malnutrition or being in risk of malnutrition is prevalent in half of the older adults receiving home care services [18]. Common consequences of a fall are fear of falling, activity restrictions, loss of mobility and loss of independence [19]. Falling, or being at risk of falling also has a negative influence on QOL [20]. Hence, it can be argued that HRQOL is an important outcome in the assessment of falls-prevention programmes [21].

After several decades of research on interventions to reduce falls and fall risk factors, there is now strong evidence for the effectiveness and cost-efficiency of exercise in reducing the number of falls [14, 22-25]. An important, but yet understudied group when it comes to the effect of falls prevention programmes are older adults receiving home help services, and especially those who recently have experienced a fall [11]. Previous research has shown that falls and fear of falling are common in this population and are correlated with the amount of home care needed [11, 26]. Vikman et al. [11] concluded that future studies should have a focus on the effects of falls prevention programmes in the group of those receiving home help services. Recently it has been shown that home help receivers fell more frequently than the independent home-dwelling older population [27]. Low functional level and high home care recipient health problems were independently associated with risk of falling [27]. Fear of falling is also reported more frequently in the group of older adults receiving home help services compared to those who do not receive home care [28]. This suggests that the higher level of fear of falling could be due to a higher level of frailty in this group. Finally, it has been shown that elderly home help receivers in Sweden have a lower QOL compared to those without help and that QOL was negatively correlated with the amount of help needed [29].

### Interventions to improve Quality of life

Although exercise-based falls prevention programmes have shown a clear effect on falls incidence and fall risk factors in the general older population, the evidence is still inconsistent about the effects on HRQOL and in particular related to the population of home help receivers [11, 21]. A systematic review by Vaapio et al. [21] considered the specific effect of falls prevention programmes on QOL. The review looked at twelve RCTs including older adults, but none of the studies were aimed at home help receivers. Six of these studies showed a positive effect on QOL. The interventions in these

studies ranged from exercise (two studies), information based (one study), to comprehensive geriatric assessment (one study). The review concluded that there is a lack of evidence about the potential benefits of falls prevention programmes on QOL in older people and that more research is needed.

To the authors' knowledge, only two RCTs have been examining exercise interventions aimed specifically at the population of older home help receivers [30, 31]. The first study tested a home-exercise programme and found positive results on maximum walking speed, but unfortunately the assessors were not blinded to the intervention [31]. The other study explored the effects and costs of a multifactorial, interdisciplinary team approach to falls prevention in 109 older home help receivers with a risk for falls [30]. Exercise was part of the programme, but the amount and mode of exercise varied according to individual needs. At six months, no difference in the mean number of falls between groups were found. Subgroup analyses showed that the intervention effectively reduced falls in men (75-84 years old) with a fear of falling or negative fall history, but it is unclear whether the study had sufficiently power for subgroup analyses [30]. Nevertheless, the secondary outcome of QOL significantly improved in the intervention group.

The effect of exercise interventions on HRQOL in the general older adult population have had mixed results, reporting both statistically significant positive effects as well as no significant changes [32-35]. A meta-analysis found no difference between aerobic and strength training, suggesting that the different exercise modes yielded the same effect on self-reported physical function domains of HRQOL [34]. Acree et al. [3] concluded that healthy older adults who regularly participated in physical activity of at least moderate intensity for more than one hour per week had higher HRQOL measures in both physical and mental domains than those who were less physically active. Although many intervention trials have found a positive association between exercise and HRQOL, the available data from other intervention trials conducted among older adults is inconsistent. Additionally, information of the most effective mode of exercise that may influence HRQOL is lacking [32-35]. Self-efficacy is a possible psychological mediating factor and physical function is a possible physiological mediating factor. Previous research has shown that self-efficacy beliefs can be related to well-being following exercise interventions [36, 37] and that self-efficacy can explain adherence to exercise programs [38-41]. A central concept of the self-efficacy theory is so-called performance accomplishment, i.e. mastery experiences related to certain activities [42], and this points towards testing the mediating effect also of physical function.

The primary aim of this study is to explore the effects of a falls prevention programme, lasting twelve weeks, on HRQOL in older adults receiving home help services. Effects on the secondary outcomes, physical function and falls efficacy, will also be explored. A secondary aim of this study is to explore the mediating factors between falls prevention and HRQOL.

# Methods

# Study design

The study is a single-blinded, pragmatic RCT comparing one intervention group with a control group. The intervention group will receive an adapted version of the Otago Exercise Programme (OEP) over twelve weeks, while the control group receives usual care. Measurements are performed at baseline, at three months and at six months. The intervention and assessments will be conducted in the participants' homes. Assessors will be blinded to group participation.

# Study setting and recruitment

Six municipalities in the Oslo region have agreed to take part in the research project. Participants are recruited through consultants in the municipalities coordinating and providing home help services. The researcher visits the municipalities on a regular basis to conduct the recruitment. Additionally, health workers in the municipalities are informed about the criteria to participate and will alert about eligible participants. Eligible participants will be contacted by the researcher by telephone and asked to consent to being sent information about the study. After a week, they will be contacted again to see if they consent orally to participate. Before baseline testing, the participants must provide a written informed consent. Figure 1 presents the planned flow of participants in the study.

#### Inclusion and exclusion criteria

Inclusion criteria are: Individuals who 1) are 67 or older, 2) receive home help services 3) have experienced at least one fall during the last twelve months, 4) are able to walk with or without a walking aid and 5) understand Norwegian. Exclusion criteria are: 1) medical contraindications to exercise, 2) life expectancy below one year, 3) a score below 23 on the Mini Mental State Examination (MMSE) and 4) currently participating in other falls prevention programmes or trials.

#### Randomisation

The participants are randomly assigned at a 1:1 ratio to the intervention group and the control group. A computer-generated, permuted block randomisation scheme is used to allocate the participants. Following randomisation, the participants receive information by telephone on which group they are allocated to. See flow chart in Figure 1.

In order to optimize the rigor of the RCT and to minimize bias, a number of methodological factors have been incorporated into the design of the study. The study participants will be randomly allocated to the groups via concealed allocation, as inadequately concealed allocation has been associated with bias in RCTs [43]. Due to the nature of the intervention, it is not possible to blind the participants or the treating therapists to the allocated groups. However, all assessors are blinded to the allocated groups. In further attempts to reduce bias, data will be analysed on an intention-to-treat basis. This preserves the randomisation process and imitate the real-life situation where the possibility exists that not all participants receive the prescribed treatment.

# Study intervention

The intervention performed is based on the OEP, including home visits and motivational phone calls [44]. Balance exercises comprise tasks in standing, walking backwards, stair-walking and rising from a chair. Strengthening exercises uses ankle weight cuffs to strengthen hip extension and abduction, knee flexion and extension and ankle plantar and dorsiflexion. The programme also includes warm-up exercises as movement of neck and shoulders. The OEP has been described in more detail previously [44]. This programme has been shown to be effective in reducing number of falls and number of injuries resulting from falls in addition to improving strength and balance, and maintaining falls efficacy in home-dwelling older adults [45].

In previous studies the OEP has been performed over a period of one year [45]. A meta-analysis by Sherrington et al. [46], looking at the effect of falls prevention programmes, recommend a dose of at least three hours of exercise weekly for six months. This weekly dose is attempted, but the duration of three months is shorter than in previous studies. Nevertheless, as in the original OEP, the same number of home visits and telephone calls will be made, and the participants will be encouraged to do a sufficient amount of exercise between home visits. The rational for the change in duration and frequency is both theoretical and pragmatic. Participants included for this study are frail older adults who have a fall history and who receive home help services. Previous research has shown that home help receivers fall more frequently and have a higher level of fear of falling [27, 47]. Poor health, fear of falling, depression and lack of strength are barriers for older adults in order to adhere to exercise programmes [48]. The participants in this study are thus likely to have a lower level of observance compared to more independent elderly and a duration of one year might be too long. Additionally, previous research has shown that falls prevention programmes which were considered too demanding by the participants even had a negative impact on QOL [49]. On the other hand, only receiving a few visits might not provide sufficient support which in turn could limit adherence. The

pragmatic rationale relates to the organizational structure of physiotherapy services in the primary health care. For this group of older adults an intervention of three months is within the time frame of what the physiotherapists normally can provide. Finally, previous research has shown that also falls prevention programmes with a shorter duration than six months have had a positive effect on QOL [21].

The physiotherapists visit the participants at home five times during the intervention (week 1, 2, 4, 8 and 10) for instruction and for guiding the appropriate level and progression of each exercise. This includes one additional visit compared to the first twelve weeks of the original OEP intervention [44]. Each visit will take about one hour. The first visit may take longer is initial information is given and a relationship is established. At this visit advice related to safety when performing exercises is provided to the participants, both orally and written. In between supervised sessions, participants will be encouraged to continue exercising on their own three times weekly for 30 minutes. Equipment for exercising (ankle cuff weights of 1, 1,5, 2 and 2,5 kg) is provided for each participant. The weeks between home visits, the physiotherapists call the participants to motivate them to continue exercising and to answer possible questions. As a part of the programme, the participants are also encouraged to perform at least two or more weekly walks of ≥30 minutes. The participants are provided with a written exercise booklet including illustrations. Following the intervention period, the participants to keep the exercise equipment and booklets, in order to continue exercising.

The participants in the control group will receive usual care from the primary health care service. Following reassessment, the participants will have opportunity to participate in other falls prevention programmes, for example, already existing balance exercise group classes.

# Education of intervention deliverers

Workshops and meetings will be held to inform the physiotherapists participating in the project. Before starting recruitment, one full day workshop on falls prevention and OEP is held for all therapists. Following start-up of recruitment and until the end of the project one workshop will be held approximately every forth months. These last half a day and include one lecture on a topic concerning older people and time for discussion on the development of the project. Additional to the workshops, the researcher will have monthly meetings with the physiotherapists in the different municipalities. In order to make sure that the intervention is performed as intended, a fidelity checklist based on the OEP-manual has been developed. The physiotherapists use the checklist when conducting the home visits and phone calls.

### Outcome measures

Following recruitment participants are assessed before they are randomised. Assessors are blinded to the participants' group assignment. The time window between baseline assessment and start of intervention is aimed to be within two weeks, and the same time window for assessments due at three and six months. Measurements and their order are selected to avoid physical and mental fatigue of the participants. Outcome measures that are employed have established reliability and validity, as recommended by the CONSORT group [50]. In addition to improving measurement quality and outcomes, it enables direct comparisons with other studies that investigate HRQOL and can possibly contribute to meta-analyses.

At baseline the Mini Mental Statement Examination (MMSE), a measurement of "Global cognitive function", is performed and is used as exclusion criteria. The maximum score is 30. A score below 23 indicates cognitive impairment and these participants are excluded [51]. Sociodemographic characteristics, like age and education, are also assessed at baseline. Primary and secondary outcome measures will be performed at baseline, at three months and at six months' follow-up.

# Primary outcome variable

HRQOL is the primary outcome measured by the Short Form 36 Health Survey (SF-36) [52]. This is a generic and validated questionnaire which, translated into Norwegian, is conducted as an interview [53]. The 36 items in SF-36 are grouped into eight health status scales: physical functioning, role limitations due to physical problems and due to emotional problems, bodily pain, general health perception, vitality, social functioning and mental health [52].

### Secondary outcome variables

In addition to the SF36, the EQ-5D (1990 EuroQOL EQ-5D) is reported. The EQ-5D is a generic and validated questionnaire [54-57]. It describes five dimensions of HRQOL (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which can take one of five responses at five levels of severity (no problems/slight problems/moderate problems/severe problems/severe problems).

Physical function includes measures of balance, gait speed, muscle strength as well as activities of daily living. The Bergs Balance Scale is a 14-item scale, which is applied to assess static and dynamic balance in older adults [58]. Gait speed is assessed by measuring usual walking speed over four meters [59] and muscle strength is measured by the 30 seconds sit to stand test [60]. Instrumental ADL is recorded using the Norwegian Version of the Lawton IADL scale, which is a valid and reliable measure of a person's self-reported ability to perform complex activities of daily living [61].

Physical activity is measured using the "Walking habits questionnaire", a valid questionnaire for walking habits and physical activity for frailer older people [62]. This questionnaire assesses general behaviour of walking, regarding how often and for how long. The following questions are asked: "Do you take a daily walk?" (yes/no) or "If you do not take a daily walk how many times per week do you take a walk?" (never/almost never/1-2 days/3-4 days/ almost daily) and "How long does you walk generally last? (0-15 mins/15-30mins/30-60mins/ 1h-2h/>2h)". Walking time in minutes per week is calculated by taking the lowest level of days multiplied by lowest level of minutes for each response alternative [62].

*Nutritional status* is measured using the Mini Nutritional Assessment (MNA- elderly, Société des Produits Nestlé, S.A., Vevey, Switzerland) form. The first screening part of six questions is used which includes measurement of weight and height for calculation of BMI [63-65].

Falls efficacy is assessed using the Falls Efficacy Scale International (FES-I). This scale has shown good reliability and validity assessing concerns about falling in older adults, and is recommended for clinical trials and practise [66, 67]. It is a self-reported questionnaire, containing 16 items on different activities of daily living. Level of concern is measured on a four-point scale ranging from 1, which is not at all concerned, to 4 which is very concerned [68].

Adherence to the programme is documented through an activity diary completed by the participants and a form checked by the physiotherapists during home visits and calls. Additionally, the participants have a falls calendar where they report adverse events. Adverse events are registered in the following four categories: falls, cardiovascular events, musculoskeletal injuries and health care utilization and will be documented as "due to the intervention" or "not due to the intervention" [69].

### Sample size estimation

The sample size is estimated from the primary outcome, HRQOL (SF-36). A treatment difference of 10 points between the two groups in one of the domains in SF-36 is regarded to be of statistical and clinical significance. The associated standard deviation is assumed to be around 20 points. This implies a moderate effect size [70], which can be expected as previous OEP studies have shown substantial effects on physical outcomes [45]. Moreover, a similar Norwegian study, which included older adults performing exercise following discharge from hospital, estimated the required sample size identically [71]. Given a power of 80% and level  $\alpha$ =0.05, we aim at including 150 participants, allowing for a 15-20% dropout, to detect a difference of 10 points between groups (see Figure 1).

# Statistical procedures

Statistical analysis is performed using SPSS or a similar statistical package. Descriptive data are reported for variables of interest. The data will be analysed following the intention to treat principle [72]. Prospective differences in primary and secondary outcomes and baseline characteristics between the intervention group and the control group will be assessed by t-tests for continuous and normal distributed variables and with non-parametric tests for categorical variables. Multiple linear regression modelling are used to control for confounding of between-group differences [73]. Hypotheses about mediating factors are tested through correlations, multiple regressions and bootstrapping methods exploring the correlations and explained variance of the chosen mediating factors and the changes in QOL [74]. Bootstrapping is a non-parametric method and is considered favourable with dichotomous variables (group 1 and 2) and small samples (n < 250) [74].

# Discussion

The main purpose of the study is to evaluate the impact of OEP on HRQOL in older adults receiving home help services. We anticipate that the intervention described in this protocol will have a positive impact on the HRQOL. The tailored intervention will have a potential to promote evidence-based decision-making and empower older people receiving home help services to remain to a greater extent in charge of their own lives. We rely on a systematic approach, which corresponds with the guidance on developing and evaluating RCTs [75]. Only a few studies have included HRQOL when measuring the effect of a falls prevention programme, and most of these studies include it as a secondary outcome [21, 76]. Outcomes examining HRQOL are selected based on literature identifying a standard set of measurements in falls prevention programmes [77, 78]. SF-36 is chosen due to its good validity, reliability and responsiveness when assessing older adults [79]. This outcome is detailed and broad, but it might be putting a burden on the participants due to its length and sensitive questions. Nevertheless, estimating HRQOL is important to determine whether the effect of a falls prevention programme is significant enough to achieve clinical relevant changes and thus to justify the implementation.

Several studies have looked at the effect of exercise on HRQOL, but to the authors' knowledge, none of them have specifically focused on older adults who receive home help services and who have a fall history. Studying the relationship between exercise and HRQOL is interesting due to the potential influence of exercise on both health and wellness through improvement of HRQOL [3, 80]. However, results from previous clinical exercise trials have reported mixed effects on HRQOL following exercise [32-35, 81]. Although many studies have found a positive association between exercise and HRQOL,

available data from other trials is inconsistent and lacks information on the most effective mode of exercise that may influence HRQOL [32, 33, 71, 81]. This study can provide insight into the effect of falls preventative exercise and its applicability to home-dwelling older fallers with dependency of help from the primary health care service.

There are two ways an intervention mechanism can influence HRQOL, it can be a mediator or a moderator [82]. A mediating factor is defined as an intervening causal factor that may provide information concerning why the intervention increases HRQOL. Moderator mechanisms help us to understand for whom an intervention works [38] and can be classified as either characteristic of the person/group i.e. baseline characteristics or characteristics of the exercise protocol [38, 83]. Mediating mechanisms between HRQOL and falls-prevention programs may be both physiological, such as increased balance and strength, and psychological, such as self-efficacy [38]. A recent study provide evidence that fear is related to falls and concluded that falls self-efficacy plays a mediation role on the relationship between fear of falls and falls [84]. They recommend that any falls prevention should consider psychological covariates of falls, especially subjects' self-efficacy to reduce falls, alongside other risk factors and covariates of falls. More theoretically driven research on these mechanisms behind treatment effects have been recommended [85-87].

It is widely accepted that falls and subsequent injuries are likely to result in a substantial reduction in quality of life for the persons affected as well a substantial economic burden to the healthcare system [88]. This provision of OEP in this setting could potentially be a beneficial and cost-effective intervention for this group of frail older adults, just as it is for community-dwelling older adults. Several studies have performed analysis on cost-effectiveness of exercise programmes which have shown that it can reduce healthcare costs [14, 89]. Due to its large sample size and theoretically based intervention the present study has the potential to generate new knowledge that may improve the design of future activity programmes for older fallers receiving home help services. Since both outcome measures as well as the intervention are carried out in a clinical setting, relevance and application of study findings to clinicians is enhanced. Results from this study will be primarily of interest to, and could be used by, health care managers and clinicians. Particularly, the results will be useful in decision making to set priorities relating to prevention measures in the community, to appropriately allocate resources and to assess costs and benefits of a falls prevention programme. Finally, the results can be useful for policy makers, in order to put preventative healthcare for this group of frail older adults on the agenda.

To conclude, older people receiving home help services represent a growing and diverse group as part of the population of community-dwelling older adults. The appropriate assessment of HRQOL, the mechanisms behind the relationship between fall prevention and HRQOL, the most effective mode of exercise, as well as the clinical relevance of the results, are challenging issues which are important to address.

# List of abbreviations

ADL Activities of Daily Living

BMI Body Mass Index

EQ-5D European Quality of Life - 5 Dimensions

HRQOL Health-related Quality of Life

iADL instrumental Activities of Daily Living

LEON lowest most efficient level of care

MMSE Mini Mental State Examination

MNA Mini Nutritional Assessment

OEP Otago Exercise Programme

pADL personal Activities of Daily Living

QOL Quality of Life

RCT Randomised Controlled Trial

SF-36 Short Form 36 Health Survey

WHO World Health Organization

# **Declarations**

# Ethics approval and consent to participate

The project proposal has been approved by The Regional Committee for Medical Research Ethics in South Norway (Ref. 2014/2051). Informed consent is obtained from all participants included in the analyses, and the project is conducted according to the WMA Declaration of Helsinki.

# Consent for publication

Not applicable

# Availability of data and materials

The datasets generated and/or analysed during the proposed study are only available to the participating researchers due to data protection laws. Subsets or aggregation of these data will not include information that could compromise research participants' privacy. Consent can be made available from the corresponding author on reasonable request.

# Competing interests

DAS is a Director of Later Life Training Ltd, a UK based non-profit organisation providing training to therapists in the effective delivery of the OEP to older adults.

# **Funding**

This study has received no external funding. It is internally funded by the Oslo and Akershus University College.

### Authors' contributions

MB and AB were involved in choosing falls prevention programme as well as outcome measures. AB was responsible for the internal grant application for this trial. MB and AB contributed to the design of the study. MB administrates the data collection and coordination of conducting the fall prevention programme. MB and AB wrote the first draft of the manuscript. TB and DAS critically revised and approved the final version of this manuscript.

### Acknowledgements

Thanks to all physiotherapists and consultants working in the municipalities contributing with information on practical issues on recruitment and management of the intervention.

## References

- 1. Luthy C, Cedraschi C, Allaz A-F, Herrmann FR, Ludwig C: **Health status and quality of life:** results from a national survey in a community-dwelling sample of elderly people. *Quality of Life Research* 2015, **24**(7):1687-1696.
- 2. Salkeld G, Ameratunga SN, Cameron I, Cumming R, Easter S, Seymour J, Kurrle S, Quine S, Brown PM: Quality of life related to fear of falling and hip fracture in older women: a time trade off studyCommentary: Older people's perspectives on life after hip fractures. *BMJ* 2000, **320**(7231):341-346.
- 3. Acree LS, Longfors J, Fjeldstad AS, Fjeldstad C, Schank B, Nickel KJ, Montgomery PS, Gardner AW: Physical activity is related to quality of life in older adults. *Health and Quality of Life Outcomes* 2006, **4**(1):1.
- 4. The WHOQOL Group: **The World Health Organization quality of life assessment (WHOQOL): development and general psychometric properties**. *Social Science & Medicine* 1998, **46**(12):1569-1585.
- 5. Helse- og omsorgsdepartementet: **NOU 2011:11. Innovasjon i omsorg.** Oslo, 2011.
- 6. Helse- og omsorgsdepartementet: **St. Meld 47. Samhandlingsreformen**. Oslo, 2009.
- 7. Christensen K, Doblhammer G, Rau R, Vaupel JW: **Ageing populations: the challenges ahead**. *The Lancet* 2009, **374**(9696):1196-1208.
- 8. Elkan R, Blair M, Robinson JJ: **Evidence-based practice and health visiting: the need for theoretical underpinnings for evaluation**. *Journal of Advanced Nursing* 2000, **31**(6):1316-1323.
- 9. Helse- og omsorgsdepartementet: **LOV-2011-06-24-30. Lov om kommunale helse- og omsorgstjenester**. Oslo, 2011.
- 10. Meinow B, Kåreholt I, Lagergren M: According to need? Predicting the amount of municipal home help allocated to elderly recipients in an urban area of Sweden. Health & Social Care in the Community 2005, 13(4):366-377.
- 11. Vikman I: Falls, perceived fall risk and activity curtailment among older people receiving home-help service. Luleå Tekniska Universitet; 2011.
- 12. Helsedirektoratet: **Prioriteringer i helsesektoren. Verdigrunnlag, status og utfordringer**. Oslo, 2012.
- 13. Vieira ER, Palmer RC, Chaves PH: **Prevention of falls in older people living in the community**. *BMJ* 2016, **353**:i1419.
- 14. Gillespie LD, Robertson MC, Gillespie WJ, Sherrington C, Gates S, Clemson LM, Lamb SE: Interventions for preventing falls in older people living in the community. *Cochrane Database Syst Rev* 2012, **9**(11).
- 15. Bergland A: **Falls suffered by the elderly living at home.** PhD thesis, University of Oslo; 2002.
- 16. Ambrose AF, Paul G, Hausdorff JM: **Risk factors for falls among older adults: a review of the literature**. *Maturitas* 2013, **75**(1):51-61.
- 17. Vivanti AP, McDonald CK, Palmer MA, Sinnott M: **Malnutrition associated with increased** risk of frail mechanical falls among older people presenting to an emergency department. *Emergency Medicine Australasia* 2009, **21**(5):386-394.
- 18. Saletti A, Johansson L, Yifter-Lindgren E, Wissing U, Österberg K, Cederholm T: **Nutritional** status and a **3-year follow-up in elderly receiving support at home**. *Gerontology* 2005, **51**(3):192-198.
- 19. Scheffer AC, Schuurmans MJ, Van Dijk N, Van Der Hooft T, De Rooij SE: **Fear of falling:** measurement strategy, prevalence, risk factors and consequences among older persons. *Age and Ageing* 2008, **37**(1):19-24.

- 20. Hawkins K, Musich S, Ozminkowski RJ, Bai M, Migliori RJ, Yeh CS: **The burden of falling on the quality of life of adults with Medicare supplement insurance**. *Journal of Gerontological Nursing* 2011, **37**(8):36-47.
- 21. Vaapio SS, Salminen MJ, Ojanlatva A, Kivelä S-L: Quality of life as an outcome of fall prevention interventions among the aged: a systematic review. *The European Journal of Public Health* 2009, **19**(1):7-15.
- 22. Campbell AJ, Robertson MC: **Rethinking individual and community fall prevention strategies: a meta-regression comparing single and multifactorial interventions**. *Age and Ageing* 2007, **36**(6):656-662.
- 23. El-Khoury F, Cassou B, Charles MA, Dargent-Molina P: The effect of fall prevention exercise programmes on fall induced injuries in community dwelling older adults: systematic review and meta-analysis of randomised controlled trials. BMJ 2013, 347:f6234.
- 24. Petridou ET, Manti EG, Ntinapogias AG, Negri E, Szczerbińska K: What works better for community-dwelling older people at risk to fall? A meta-analysis of multifactorial versus physical exercise-alone interventions. *Journal of Aging and Health* 2009, **21**(5):713-729.
- 25. Sherrington C, Whitney JC, Lord SR, Herbert RD, Cumming RG, Close JC: **Effective exercise for the prevention of falls: a systematic review and meta-analysis**. *Journal of the American Geriatrics Society* 2008, **56**(12):2234-2243.
- 26. Vikman I, Nordlund A, Näslund A, Nyberg L: **Incidence and seasonality of falls amongst old people receiving home help services in a municipality in northern Sweden**. *International Journal of Circumpolar Health* 2011, **70**(2):195.
- 27. Meyer C, Dow B, Bilney BE, Moore KJ, Bingham AL, Hill KD: Falls in older people receiving inhome informal care across Victoria: Influence on care recipients and caregivers.

  Australasian Journal on Ageing 2012, 31(1):6-12.
- 28. Fletcher PC, Hirdes JP: **Restriction in activity associated with fear of falling among community-based seniors using home care services**. *Age and Ageing* 2004, **33**(3):273-279.
- 29. Hellström Y, Persson G, Hallberg IR: **Quality of life and symptoms among older people living at home**. *Journal of Advanced Nursing* 2004, **48**(6):584-593.
- 30. Markle-Reid M, Browne G, Gafni A, Roberts J, Weir R, Thabane L, Miles M, Vaitonis V, Hecimovich C, Baxter P: **The effects and costs of a multifactorial and interdisciplinary team approach to falls prevention for older home care clients 'at risk'for falling: a randomized controlled trial**. *Canadian Journal on Aging 2010*, **29**(01):139-161.
- 31. Bonnefoy M, Boutitie F, Mercier C, Gueyffier F, Carre C, Guetemme G, Ravis B, Laville M, Cornu C: Efficacy of a home-based intervention programme on the physical activity level and functional ability of older people using domestic services: a randomised study. The Journal of Nutrition, Health & Aging 2012, 16(4):370-377.
- 32. Chou C-H, Hwang C-L, Wu Y-T: Effect of exercise on physical function, daily living activities, and quality of life in the frail older adults: a meta-analysis. *Archives of Physical Medicine and Rehabilitation* 2012, **93**(2):237-244.
- 33. Gillison FB, Skevington SM, Sato A, Standage M, Evangelidou S: **The effects of exercise** interventions on quality of life in clinical and healthy populations; a meta-analysis. *Social Science & Medicine* 2009, **68**(9):1700-1710.
- 34. Kelley GA, Kelley KS, Hootman JM, Jones DL: Exercise and health-related quality of life in older community-dwelling adults a meta-analysis of randomized controlled trials. *Journal of Applied Gerontology* 2009, **28**(3):369-394.
- 35. De Vries N, Van Ravensberg C, Hobbelen J, Rikkert MO, Staal J, Nijhuis-van der Sanden M: Effects of physical exercise therapy on mobility, physical functioning, physical activity and quality of life in community-dwelling older adults with impaired mobility, physical disability and/or multi-morbidity: a meta-analysis. *Ageing Research Reviews* 2012, 11(1):136-149.

- 36. White SM, Wójcicki TR, McAuley E: **Physical activity and quality of life in community dwelling older adults**. *Health and Quality of Life Outcomes* 2009, **7**(1):1.
- 37. McAuley E, Konopack JF, Morris KS, Motl RW, Hu L, Doerksen SE, Rosengren K: **Physical** activity and functional limitations in older women: influence of self-efficacy. *The Journals of Gerontology Series B: Psychological Sciences and Social Sciences* 2006, **61**(5):P270-P277.
- 38. Kraemer HC, Wilson GT, Fairburn CG, Agras WS: **Mediators and moderators of treatment effects in randomized clinical trials**. *Archives of General Psychiatry* 2002, **59**(10):877-883.
- 39. McAuley E, Lox C, Duncan TE: **Long-term maintenance of exercise, self-efficacy, and physiological change in older adults**. *Journal of Gerontology* 1993, **48**(4):P218-P224.
- 40. McAuley E, Jerome GJ, Marquez DX, Elavsky S, Blissmer B: Exercise self-efficacy in older adults: social, affective, and behavioral influences. *Annals of Behavioral Medicine* 2003, **25**(1):1-7.
- 41. Landers DM, SM A: Physical activity and mental health. Hoboken, New Jersey: Wiley; 2007.
- 42. Bandura A: **Self efficacy: the exercise of control**. New York: W.H. Freeman; 1997.
- 43. Schulz KF, Chalmers I, Hayes RJ, Altman DG: **Empirical evidence of bias: dimensions of methodological quality associated with estimates of treatment effects in controlled trials**. *Jama* 1995, **273**(5):408-412.
- 44. Campbell AJ, Robertson C: **Otago Exercise programme to prevent falls in older adults**. In. Edited by School OM. Otago; 2003.
- 45. Robertson MC, Campbell AJ, Gardner MM, Devlin N: **Preventing injuries in older people by preventing falls: A meta-analysis of individual-level data**. *Journal of the American Geriatrics Society* 2002, **50**(5):905-911.
- 46. Sherrington C, Michaleff ZA, Fairhall N, Paul SS, Tiedemann A, Whitney J, Cumming RG, Herbert RD, Close JC, Lord SR: Exercise to prevent falls in older adults: an updated systematic review and meta-analysis. *British Journal of Sports Medicine* 2016:bjsports-2016-096547.
- 47. Fletcher PC, Hirdes JP: **Risk factors for falling among community-based seniors using home care services**. *The Journals of Gerontology Series A: Biological Sciences and Medical Sciences* 2002, **57**(8):M504-M510.
- 48. Forkan R, Pumper B, Smyth N, Wirkkala H, Ciol MA, Shumway-Cook A: **Exercise adherence following physical therapy intervention in older adults with impaired balance**. *Physical Therapy* 2006, **86**(3):401-410.
- 49. Vaapio S, Salminen M, Vahlberg T, Sjösten N, Isoaho R, Aarnio P, Kivelä S-L: **Effects of risk-based multifactorial fall prevention on health-related quality of life among the community-dwelling aged: a randomized controlled trial**. *Health and Quality of Life Outcomes* 2007, **5**(1):1.
- 50. Schulz KF, Altman DG, Moher D: **CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials**. *BMC Medicine* 2010, **8**(1):1.
- 51. Tombaugh TN, McIntyre NJ: **The mini-mental state examination: a comprehensive review**. *Journal of the American Geriatrics Society* 1992, **40**(9):922-935.
- 52. Ware Jr JE, Sherbourne CD: **The MOS 36-item short-form health survey (SF-36): I. Conceptual framework and item selection**. *Medical Care* 1992:473-483.
- 53. Loge JH, Kaasa S: **Short form 36 (SF-36) health survey: normative data from the general Norwegian population**. *Scandinavian Journal of Public Health* 1998, **26**(4):250-258.
- 54. The EuroQol Group: **EuroQol-a new facility for the measurement of health-related quality of life**. *Health policy* 1990, **16**(3):199-208.
- 55. Brooks R, Group E: **EuroQol: the current state of play**. *Health Policy* 1996, **37**(1):53-72.
- 56. Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X: **Development** and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Quality of Life Research 2011, **20**(10):1727-1736.

- 57. Janssen M, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J: Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. *Quality of Life Research* 2013, **22**(7):1717-1727.
- 58. Berg KO, Maki BE, Williams JI, Holliday PJ, Wood-Dauphinee SL: **Clinical and laboratory measures of postural balance in an elderly population**. *Archives of Physical Medicine and Rehabilitation* 1992, **73**(11):1073-1080.
- 59. Peters DM, Fritz SL, Krotish DE: **Assessing the reliability and validity of a shorter walk test compared with the 10-meter walk test for measurements of gait speed in healthy, older adults**. *Journal of Geriatric Physical Therapy* 2013, **36**(1):24-30.
- 60. Jones CJ, Rikli RE, Beam WC: A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Research Quarterly for Exercise and Sport 1999, 70(2):113-119.
- 61. Lawton M, Brody E: **Assessment of older people: self-maintaining and instrumental activities of daily living**. *Nursing Research* 1970, **19**(3):278.
- 62. Frändin K, Grimby G, Mellström D, Svanborg A: **Walking habits and health-related factors in a 70-year-old population**. *Gerontology* 1991, **37**(5):281-288.
- 63. Vellas B, Villars H, Abellan G, Soto M: **Overview of the MNA® Its history and challenges**. *The Journal of Nutrition, Health & Aging* 2006, **10**(6):456.
- 64. Rubenstein LZ, Harker JO, Salvà A, Guigoz Y, Vellas B: Screening for undernutrition in geriatric practice developing the short-form mini-nutritional assessment (MNA-SF). The Journals of Gerontology Series A: Biological Sciences and Medical Sciences 2001, 56(6):M366-M372.
- 65. Guigoz Y, Jensen G, Thomas D, Vellas B: **The mini nutritional assessment (MNA®). Review of the literature What does it tell us?** *The Journal of Nutrition, Health & Aging* 2006, **10**(6):466.
- 66. Delbaere K, Close JC, Mikolaizak AS, Sachdev PS, Brodaty H, Lord SR: **The falls efficacy scale international (FES-I). A comprehensive longitudinal validation study**. *Age and Ageing* 2010, **39**(2):210-216.
- 67. Marques-Vieira CMA, Sousa LMM, Severino S, Sousa L, Caldeira S: **Cross-cultural validation of the falls efficacy scale international in elderly: Systematic literature review**. *Journal of Clinical Gerontology and Geriatrics* 2016, **7**(3):72-76.
- 68. Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C: **Development and initial** validation of the Falls Efficacy Scale-International (FES-I). Age and Ageing 2005, **34**(6):614-619.
- 69. Ory M, Resnick B, Jordan PJ, Coday M, Riebe D, Garber CE, Pruitt L, Bazzarre T: **Screening**, safety, and adverse events in physical activity interventions: collaborative experiences from the behavior change consortium. *Annals of Behavioral Medicine* 2005, **29**(2):20-28.
- 70. Cohen, J: A power primer *Psychological Bulletin*, **112**(1):155-159.
- 71. Brovold T, Skelton DA, Bergland A: Older Adults Recently Discharged from the Hospital: Effect of Aerobic Interval Exercise on Health-Related Quality of Life, Physical Fitness, and Physical Activity. *Journal of the American Geriatrics Society* 2013, **61**(9):1580-1585.
- 72. Hollis S, Campbell F: **What is meant by intention to treat analysis? Survey of published randomised controlled trials**. *BMJ* 1999, **319**(7211):670-674.
- 73. Altman D: Practical statistics for medical research. London: Chapman and Hall; 1991.
- 74. Preacher KJ, Hayes AF: **Asymptotic and resampling strategies for assessing and comparing indirect effects in multiple mediator models**. *Behavior Research Methods* 2008, **40**(3):879-891.
- 75. Senn B, Kirsch M, Sanz C, Karlou C, Tulus K, De Leeuw J, Ringner A: **Developing and evaluating complex interventions: the new Medical Research Council guidance**. *Studies* 2013, **59**:587-592.

- 76. McInnes E, Askie L: Evidence review on older people's views and experiences of falls prevention strategies. Worldviews Evidence Based Nursing 2004, 1(1):20-37.
- 77. Lamb SE, Jørstad-Stein EC, Hauer K, Becker C: **Development of a common outcome data set for fall injury prevention trials: the Prevention of Falls Network Europe consensus**. *Journal of the American Geriatrics Society* 2005, **53**(9):1618-1622.
- 78. Lamb SE, Becker C, Gillespie LD, Smith JL, Finnegan S, Potter R, Pfeiffer K: **Reporting of complex interventions in clinical trials: development of a taxonomy to classify and describe fall-prevention interventions**. *Trials* 2011, **12**(1):1.
- 79. Haywood K, Garratt A, Fitzpatrick R: **Quality of life in older people: a structured review of generic self-assessed health instruments**. *Quality of Life Research* 2005, **14**(7):1651-1668.
- 80. Vuillemin A, Boini S, Bertrais S, Tessier S, Oppert J-M, Hercberg S, Guillemin F, Briançon S: Leisure time physical activity and health-related quality of life. *Preventive Medicine* 2005, 41(2):562-569.
- 81. Heydarnejad S, Dehkordi AH: **The effect of an exercise program on the health-quality of life in older adults**. *Danish Medical Bulletin* 2010, **57**(4):113-117.
- 82. Michie S, Abraham C: Interventions to change health behaviours: evidence-based or evidence-inspired? *Psychology & Health* 2004, **19**(1):29-49.
- 83. Solberg PA: Exercise and well-being among older adults: A self-determination theory perspective. PhD thesis, Norwegian School of Sports Science 2013.
- 84. Dadgari A, Hamid TA, Hakim MN, Mousavi SA, Dadvar L, Mohammadi M, Amerian N: **The role** of self-efficacy on fear of falls and fall among elderly community dwellers in Shahroud, Iran. *Nursing Practice Today* 2016, **2**(3):112-120.
- 85. McAuley E, Blissmer B, Katula J, Duncan TE: Exercise environment, self-efficacy, and affective responses to acute exercise in older adults. *Psychology and Health* 2000, **15**(3):341-355.
- 86. Netz Y, Wu M-J, Becker BJ, Tenenbaum G: Physical activity and psychological well-being in advanced age: a meta-analysis of intervention studies. *Psychology and Aging* 2005, **20**(2):272.
- 87. Standage M, JL D: **Motivational responses among older adults in sport and exercise settings**. *I: Weiss MR (red) Developmental sport and exercise psychology A lifespan perspective* 2004:357-381.
- 88. World Health Organization: **WHO Global Report on Falls Prevention in Older Age**. Geneva, 2007.
- 89. Hektoen LF, Aas E, Lurås H: **Cost-effectiveness in fall prevention for older women**. *Scandinavian Journal of Public Health* 2009, **37**(6):584-589.



Figure 1: Planned flow of participants in the study.



SPIRIT 2013 Checklist: Recommended items to address in a clinical trial protocol and related documents\*

| Section/item | Item<br>No | Description | Addressed on page number |
|---|---|---|---|
| Administrative inf | ormatio | n | |
| Title | 1 | Descriptive title identifying the study design, population, interventions, and, if applicable, trial acronym | 1, 2 |
| Trial registration | 2a | Trial identifier and registry name. If not yet registered, name of intended registry | 2 |
| | 2b | All items from the World Health Organization Trial Registration Data Set | 2 |
| Protocol version | 3 | Date and version identifier | |
| Funding | 4 | Sources and types of financial, material, and other support | 14 |
| Roles and responsibilities | 5a | Names, affiliations, and roles of protocol contributors | 1, 14 |
| | 5b | Name and contact information for the trial sponsor | 14 |
| | 5c | Role of study sponsor and funders, if any, in study design; collection, management, analysis, and interpretation of data; writing of the report; and the decision to submit the report for publication, including whether they will have ultimate authority over any of these activities | 14 |
| | 5d | Composition, roles, and responsibilities of the coordinating centre, steering committee, endpoint adjudication committee, data management team, and other individuals or groups overseeing the trial, if applicable (see Item 21a for data monitoring committee) | 14 |

# Introduction

| Background and rationale | 6a | Description of research question and justification for undertaking the trial, including summary of relevant studies (published and unpublished) examining benefits and harms for each intervention | 3-5 |
|---|---|---|---|
| | 6b | Explanation for choice of comparators | 6 |
| Objectives | 7 | Specific objectives or hypotheses | 5, 10-11 |
| Trial design | 8 | Description of trial design including type of trial (eg, parallel group, crossover, factorial, single group), allocation ratio, and framework (eg, superiority, equivalence, noninferiority, exploratory) | 6 |
| Methods: Participa | nts, int | erventions, and outcomes | |
| Study setting | 9 | Description of study settings (eg, community clinic, academic hospital) and list of countries where data will be collected. Reference to where list of study sites can be obtained | 6 |
| Eligibility criteria | 10 | Inclusion and exclusion criteria for participants. If applicable, eligibility criteria for study centres and individuals who will perform the interventions (eg, surgeons, psychotherapists) | 6 |
| Interventions | 11a | Interventions for each group with sufficient detail to allow replication, including how and when they will be administered | 7-8 |
| | 11b | Criteria for discontinuing or modifying allocated interventions for a given trial participant (eg, drug dose change in response to harms, participant request, or improving/worsening disease) | |
| | 11c | Strategies to improve adherence to intervention protocols, and any procedures for monitoring adherence (eg, drug tablet return, laboratory tests) | 8, 10 |
| | 11d | Relevant concomitant care and interventions that are permitted or prohibited during the trial | 6 |
| Outcomes | 12 | Primary, secondary, and other outcomes, including the specific measurement variable (eg, systolic blood pressure), analysis metric (eg, change from baseline, final value, time to event), method of aggregation (eg, median, proportion), and time point for each outcome. Explanation of the clinical relevance of chosen efficacy and harm outcomes is strongly recommended | 8-10 |
| Participant timeline | 13 | Time schedule of enrolment, interventions (including any run-ins and washouts), assessments, and visits for participants. A schematic diagram is highly recommended (see Figure) | 6-7, 9, Figure 1 |

| Sample size | 14 | Estimated number of participants needed to achieve study objectives and how it was determined, including clinical and statistical assumptions supporting any sample size calculations | 10 |
|---|---|---|---|
| Recruitment | 15 | Strategies for achieving adequate participant enrolment to reach target sample size | 6 |
| Methods: Assignm | ent of i | nterventions (for controlled trials) | |
| Allocation: | | | |
| Sequence<br>generation | 16a | Method of generating the allocation sequence (eg, computer-generated random numbers), and list of any factors for stratification. To reduce predictability of a random sequence, details of any planned restriction (eg, blocking) should be provided in a separate document that is unavailable to those who enrol participants or assign interventions | 6-7 |
| Allocation concealment mechanism | 16b | Mechanism of implementing the allocation sequence (eg, central telephone; sequentially numbered, opaque, sealed envelopes), describing any steps to conceal the sequence until interventions are assigned | 6-7, |
| Implementation | 16c | Who will generate the allocation sequence, who will enrol participants, and who will assign participants to interventions | 6 |
| Blinding (masking) | 17a | Who will be blinded after assignment to interventions (eg, trial participants, care providers, outcome assessors, data analysts), and how | 7-9 |
| | 17b | If blinded, circumstances under which unblinding is permissible, and procedure for revealing a participant's allocated intervention during the trial | 6 |
| Methods: Data collection, management, and analysis | | | |
| Data collection methods | 18a | Plans for assessment and collection of outcome, baseline, and other trial data, including any related processes to promote data quality (eg, duplicate measurements, training of assessors) and a description of study instruments (eg, questionnaires, laboratory tests) along with their reliability and validity, if known. Reference to where data collection forms can be found, if not in the protocol | 8-10 |
| | 18b | Plans to promote participant retention and complete follow-up, including list of any outcome data to be collected for participants who discontinue or deviate from intervention protocols | 7 |

| Data management | 19 | Plans for data entry, coding, security, and storage, including any related processes to promote data quality (eg, double data entry; range checks for data values). Reference to where details of data management procedures can be found, if not in the protocol | Included in ethical approval, p.14 |
|---|---|---|---|
| Statistical methods | 20a | Statistical methods for analysing primary and secondary outcomes. Reference to where other details of the statistical analysis plan can be found, if not in the protocol | 10 |
| | 20b | Methods for any additional analyses (eg, subgroup and adjusted analyses) | 10 |
| | 20c | Definition of analysis population relating to protocol non-adherence (eg, as randomised analysis), and any statistical methods to handle missing data (eg, multiple imputation) | 6-7 |
| Methods: Monitorii | Methods: Monitoring | | |
| Data monitoring | 21a | Composition of data monitoring committee (DMC); summary of its role and reporting structure; statement of whether it is independent from the sponsor and competing interests; and reference to where further details about its charter can be found, if not in the protocol. Alternatively, an explanation of why a DMC is not needed | 14 |
| | 21b | Description of any interim analyses and stopping guidelines, including who will have access to these interim results and make the final decision to terminate the trial | 10, 14 |
| Harms | 22 | Plans for collecting, assessing, reporting, and managing solicited and spontaneously reported adverse events and other unintended effects of trial interventions or trial conduct | 10 |
| Auditing | 23 | Frequency and procedures for auditing trial conduct, if any, and whether the process will be independent from investigators and the sponsor | NA |
| Ethics and dissemination | | | |
| Research ethics approval | 24 | Plans for seeking research ethics committee/institutional review board (REC/IRB) approval | 14 |
| Protocol amendments | 25 | Plans for communicating important protocol modifications (eg, changes to eligibility criteria, outcomes, analyses) to relevant parties (eg, investigators, REC/IRBs, trial participants, trial registries, journals, regulators) | 14 |

| Consent or assent | 26a | Who will obtain informed consent or assent from potential trial participants or authorised surrogates, and how (see Item 32) | 6, 14 |
|---|---|---|---|
| | 26b | Additional consent provisions for collection and use of participant data and biological specimens in ancillary studies, if applicable | NA |
| Confidentiality | 27 | How personal information about potential and enrolled participants will be collected, shared, and maintained in order to protect confidentiality before, during, and after the trial | Included in ethical approval, p.14 |
| Declaration of interests | 28 | Financial and other competing interests for principal investigators for the overall trial and each study site | 14 |
| Access to data | 29 | Statement of who will have access to the final trial dataset, and disclosure of contractual agreements that limit such access for investigators | 14 |
| Ancillary and post-<br>trial care | 30 | Provisions, if any, for ancillary and post-trial care, and for compensation to those who suffer harm from trial participation | 8 |
| Dissemination policy | 31a | Plans for investigators and sponsor to communicate trial results to participants, healthcare professionals, the public, and other relevant groups (eg, via publication, reporting in results databases, or other data sharing arrangements), including any publication restrictions | 14 |
| | 31b | Authorship eligibility guidelines and any intended use of professional writers | |
| | 31c | Plans, if any, for granting public access to the full protocol, participant-level dataset, and statistical code | 14 |
| Appendices | | | |
| Informed consent materials | 32 | Model consent form and other related documentation given to participants and authorised surrogates | Included in ethical approval |
| Biological specimens | 33 | Plans for collection, laboratory evaluation, and storage of biological specimens for genetic or molecular analysis in the current trial and for future use in ancillary studies, if applicable | |

<sup>\*</sup>It is strongly recommended that this checklist be read in conjunction with the SPIRIT 2013 Explanation & Elaboration for important clarification on the items. Amendments to the protocol should be tracked and dated. The SPIRIT checklist is copyrighted by the SPIRIT Group under the Creative Commons "Attribution-NonCommercial-NoDerivs 3.0 Unported" license.